CLINICAL TRIAL: NCT02203045
Title: Outcomes Following Tourniquet and Non-Tourniquet Assisted Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Joint Replacement (Other); CommonSpirit Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-0648
Record Dates: First submitted 2014-07-24; First posted 2014-07-29 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2014-10

CONDITIONS: Osteoarthritis
Keywords: Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tourniquet (Active Comparator): All lower extremities will be exsanguinated by elevation for 2 minutes. For lower extremities in the tourniquet group (TQT), a pneumatic tourniquet will be inflated according to standard practice (>200 mmHg). For the NOTQT group, the tourniquet will only be inflated during component cementation. In both groups, tourniquet will be deflated after bone cement has set. In both groups, electrocautery will be used as needed throughout the procedure.
  Interventions: Other: Total Knee Arthroplasty
- Non- tourniquet (Experimental): All lower extremities will be exsanguinated by elevation for 2 minutes. For lower extremities in the tourniquet group (TQT), a pneumatic tourniquet will be inflated according to standard practice (>200 mmHg). For the NOTQT group, the tourniquet will only be inflated during component cementation. In both groups, tourniquet will be deflated after bone cement has set. In both groups, electrocautery will be used as needed throughout the procedure.
  Interventions: Other: Total Knee Arthroplasty

INTERVENTIONS:
Other: Total Knee Arthroplasty

SUMMARY:
The overall goal of this study is to determine the effects of intraoperative tourniquet use during total knee arthroplasty (TKA), compared to TKA without the use of a tourniquet (NOTQT), for strength and functional recovery following simultaneous bilateral TKA. During the procedure, each patient will receive tourniquet-assisted TKA (TQT) on one lower extremity while the contralateral lower extremity undergoes TKA without the use of a tourniquet (NOTQT), except for briefly during component cementation. Tourniquets are commonly used in TKA to improve visualization of the surgical field and limit blood loss. However, studies suggest that tourniquet use may be associated with higher rates of medical complications and poor functional outcomes, including increased swelling, decreased muscle strength and altered neuromuscular activity. We will measure strength, voluntary muscle activation, and other functional outcomes for each lower extremity at 4 time points (preop; inpatient (24-72 hrs after surgery); 3 weeks; and 3 months following TKA). We hypothesize that lower extremities in the NOTQT group will demonstrate improved strength and performance when compared to lower extremities in the TQT group.

ELIGIBILITY:
Inclusion Criteria:

* undergoing primary, simultaneous bilateral knee arthroplasty for osteoarthritis

Exclusion Criteria:

* no neurological, vascular or cardiac problems that limit function or any unstable orthopaedic conditions that limit functional performance

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-10; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Quadriceps Muscle Force | Pre-operative, 3 weeks and 3 months post-operative
  NOTQT will result in greater quadriceps muscle strength (primary outcome) after TKA, compared to TQT group. Benefits will be apparent at 48-72 hrs and 3 weeks (primary endpoint), and persist though 3 months following TKA

SECONDARY OUTCOMES:
Change from Baseline in Balance testing | Pre-operatively, 3 weeks and 3 months post-operative
  Patients will be asked to perform a test of unilateral balance ability. Patients will place both hands on their hips before assuming a single limb stance. Patients will attempt to hold this position for a maximum time of 60 seconds, although timing will stop if patients ever place both feet on the ground, if the non-stance leg braces against the stance leg to control balance, or if hands are removed from the hips to regain balance.
Change from Baseline in Isometric Hamstring Strength | Pre-operatively, 3 weeks and 3 months post-operative
Change from Baseline from Voluntary Quadriceps Activation | Pre-operative, 3 weeks and 3 months post-operative
Change from Baseline in Range of Motion | Pre-operatively, 3 weeks and 3 months post-operatively
  Knee flexion and extension range of motion (ROM) will be quantified using a standard long-arm goniometer with the patient lying in supine. Knee flexion ROM will be defined as the angle of maximal active bending of the knee. Knee extension ROM will be the angle of maximal straightening while the patient's heel is propped on a 10cm wooden block. If hyperextension is achieved, then the degrees of extension beyond zero will be recorded as a negative value.

OTHER OUTCOMES:
Radiographic Examination | 1 to 2 months post surgery
  Radiographic examination will be used to provide preliminary data on rates of fracture and tibiofemoral joint malalignment specific to the use of tourniquet during surgery.
Deep Vein Thrombosis Formation | 48- 72 hours post operative
Postoperative blood loss | 48 hours post surgery
Lower extremity edema | 48- 72 hours postoperative
Verbal analog scale pain assessment | Pre-Operative, 3 weeks and 3 months post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Dennis, MD, Principal Investigator — Colorado Joint Replacement; Jennifer Stevens-Lapsley, MPT and PhD, Study Director — University of Colorado, Denver; Ray Kim, MD, Principal Investigator — Colorado Joint Replacement
Locations (2):
- United States (2):
  - Univeristy of Colorado, Aurora, Colorado
  - Colorado Joint Replacement, Denver, Colorado